CLINICAL TRIAL: NCT06414850
Title: Efficacy Study of an Animal-assisted Intervention in Adolescents Admitted to Acute Psychiatric Units: Mentaldog Multicenter Study.
Brief Title: Animal-assisted Intervention in Adolescents Admitted to Acute Psychiatric Units.
Acronym: MENTAL-DOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Hospital Universitari Santa Maria, Lleida (Unknown); Hospital de Mataró (Other); Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other); Universidad Rey Juan Carlos (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: Multicenter study
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Mental Health Issue
Keywords: Animal-assisted therapy; Mental Health; Adolescent Psychiatry; Hospital; Nonpharmaceutical interventions
MeSH Terms: conditions — Psychological Well-Being | interventions — Animal Assisted Therapy

STUDY DESIGN:
Intervention Model Description: Multicenter, non-randomized, controlled, open-label, two-arm clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (EG) (Experimental): The experimental group carried out a total of two one-hour group sessions at the three hospitals' own facilities, on a weekly basis for two consecutive weeks. The groups were formed by 8-10 participants. Sessions included the participation of one certified therapy dog, one technician specialized in AAT, an occupational therapist and a psychologist. There was a referring psychiatrist for the project at each center. Participants received their usual pharmacological treatment.
  Intervention (with the additional assistance of the therapy dog): Session 1, self-efficacy (executive functions, cause-effect thinking). Session 2, emotional self-regulation and frustration tolerance.
  Interventions: Behavioral: Animal Assisted Therapy (AAT)
- Control Group (CG) (Active Comparator): The control group carried out a total of two one-hour group sessions at the hospital's own facility, on a weekly basis for two consecutive weeks. The groups were formed by 8-10 participants. Sessions included the participation of an occupational therapist and a psychologist. There was a referring psychiatrist for the project. Participants received their usual pharmacological treatment.
  Intervention (same sessions without the therapy dog): Session 1, self-efficacy (executive functions, cause-effect thinking). Session 2, emotional self-regulation and frustration tolerance.
  Interventions: Behavioral: Animal Assisted Therapy (AAT)

INTERVENTIONS:
Behavioral: Animal Assisted Therapy (AAT) — A structured AAT program and pharmacological treatment in Experimental group. The same structured program without therapy dog and pharmacological treatment in Control group.
  Other Names: Dog assisted Therapy

SUMMARY:
The purpose of the present study was to evaluate the efficacy of AAT intervention in adolescents admitted to the Acute Child and Adolescent Psychiatry Unit, regardless of diagnosis, in terms of improving self-efficacy and reducing anxiety symptoms. To assess professional opinions on the effects of intervention on participants, and to determine participant satisfaction. These objectives were accomplished through a multicenter, non-randomized, open-label, two-arm controlled study of AAT for adolescents with mental disorders.

DETAILED DESCRIPTION:
The rationale of this study was to evaluate the efficacy of Animal Assisted Therapy (with therapy dogs) in adolescents admitted to the Acute Child and Adolescent Psychiatry Unit and regardless of diagnosis. The investigators conducted a multicenter, non-randomized, controlled, open-label, two-arm clinical trial in three hospitals. A total of 178 adolescents admitted to the Acute Child and Adolescent Psychiatry Unit were included in the study. Participants from the three hospitals were assigned to Experimental Group (n=114) and participants from one hospital were assigned to Control Group (n=64). Both the experimental group and the control group carried out a total of two one-hour group sessions at the hospitals' own facilities, on a weekly basis for two consecutive weeks; with the additional assistance of the therapy dog in the Experimental group. The investigators evaluated changes on self-efficacy and anxiety symptoms at pre-treatment and post-treatment; and they assessed professional opinions on the effects of intervention on participants at post-treatment, and determined participant satisfaction at post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Be between 13 and 17 years of age.
* Willing to participate in the study on a voluntary basis.
* Delivery of the information sheet and signature of the informed consent (participant and legal guardian).
* Attendance at both group sessions from the intervention.

Exclusion Criteria:

* If in the initial interview they declared having allergy or fear of dogs.
* History of aggression towards animals.
* Re-admissions who had already participated in the study.
* If, when informed, the patient and/or his/her legal guardian did not wish to participate in the study.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 178 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline General Self-Efficacy Scale (GSE) at 2 weeks. | This scale was administered at baseline and at week 2
  Is a generic self-administered instrument for measuring self-efficacy beliefs in certain life situations. The total scale score ranges from 10 to 40 points.
Change from baseline State-Trait Anxiety Inventory Questionnaire (STAI) at 2 weeks. | This questionnaire was administered at baseline and at week 2
  Is a self-administered questionnaire that assesses the levels of clinical anxiety (both trait anxiety ("most of the time") and state anxiety ("at the present moment")). The total score on each of the subscales ranges from 0 to 60 points.

SECONDARY OUTCOMES:
Participant evaluation questionnaire for professionals. | At the end of the intervention (week 2).
  This is a questionnaire that was completed by the professionals in the three hospitals at the end of the intervention with the EG, using a Likert scale from 1 to 4 (1= Not at all, 2= Somewhat, 3= Quite, and 4= A lot). It contains the following questions:
  * Have you observed any positive changes in the patient's attitude since the AAT session?
  * Has the dog generated motivation?
  * Do you consider AAT useful for this patient?

OTHER OUTCOMES:
Participant satisfaction questionnaire at the end of the intervention. | At the end of the intervention (week 2).
  The following question was asked in writing and answered by all participants (CG + EG): Did you enjoy the activity that was carried out? It consists of a Likert scale of 1= Not at all, 2= Somewhat, 3= Quite and 4= A lot.

CONTACTS AND LOCATIONS:
Overall Officials: M. Dolores Rodrigo Claverol, PhD, Principal Investigator — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Locations (3):
- Spain (3):
  - Hospital de Mataró, Mataró, Barcelona
  - Hospital Universitari Santa Maria, Lleida
  - Hospital Universitario Infantil Niño Jesús, Madrid

IPD SHARING:
Plan to Share IPD: No